CLINICAL TRIAL: NCT03968250
Title: Cognitive Behavioral Therapy (CBT) Web-based Intervention on Fatigue in Survivors of Hodgkin Lymphoma - a Pilot Study
Brief Title: CBT on Fatigue in Survivors of Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Deutsche José Carreras Leukämie-Stiftung e.V. (Germany) (Unknown); Medical University of Cologne (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Head of the Department of Medical Psychology and Medical Sociology, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 933 000-146
Record Dates: First submitted 2018-08-24; First posted 2019-05-30 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hodgkin Lymphoma; Fatigue
MeSH Terms: conditions — Hodgkin Disease; Fatigue | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The design of this pilot web-based CBT Fatigue therapy will be a non-randomised prospective non-controlled before-and-after study, in which observations will be made only in a patient group that receives the intervention (IG). No control group will be recruited. Assessments will be conducted at three measurement points: T0 (before the intervention), T1 (at the end of the intervention), T2 (3 months after T1).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy for Treating Fatigue (Experimental): This is the patient group that receives the intervention (IG), i.e., the cognitive behavioral therapy for reducing fatigue.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Treating Fatigue

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Treating Fatigue — The internet-based CBT postcancer fatigue intervention includes two face-to-face sessions with their therapist and eight web-based treatment modules, each approximately 45 minutes in length, delivered over 6 months.
  The intervention will be specifically tailored to the individual needs of each patient: The CBT model of cancer-related fatigue distinguishes six perpetuating factors: 1) insufficient processing of being diagnosed with HL and being treated for it; 2) excessive fear of disease recurrence; 3) inactivity or a dysregulated (physical) activity pattern; 4) dysfunctional fatigue-related beliefs; 5) dysregulated sleep-wake pattern and 6) lack of social support. For each of these six cognitive-behavioural factors that can perpetuate fatigue a treatment module has been developed.

SUMMARY:
Background: Cancer-related fatigue is one of the most common patient-reported impairments in survivors of Hodgkin lymphoma and is associated with adverse effects on psychological well-being and everyday life including family, work and social participation.

Methods: The investigators here present a bi-centric (Cologne and Leipzig) pilot-study for a web-based intervention (Cognitive Behavioral Therapy) on cancer-related fatigue. In detail, the investigators will conduct a non-randomized and non-controlled before-and-after study in a minimum of 20 survivors of Hodgkin lymphoma. Levels of fatigue and quality of life will be measured before the intervention (T0), post-intervention (T1) and at 3-months follow-up (T2).

Results: The investigators will provide information regarding the feasibility of the intervention (i.e., response rate, patient and therapist adherence, and patient satisfaction) and preliminary results on the efficacy of the program in reducing CRF and increasing levels of quality of life.

Aims: The results of this pilot-study will provide essential information to conduct a future randomized clinical trial to investigate the efficacy of this intervention in reducing cancer-related fatigue in survivors with Hodgkin lymphoma.

DETAILED DESCRIPTION:
Concrete Aims: The investigators aim to conduct a a feasibility study, e.g., a pilot study before a randomized controlled trial can be planned in detail. This initial pilot-study is intended to test out the standard operating procedures, evaluate the feasibility, acceptance and adherence to the study protocol as well as preliminary efficacy of the web-based intervention for survivors of Hodgkin lymphoma. In detail, this study contains all preparation for conducting a trial, i.e., the translation, the adaptation and evaluation of the cognitive-behavioral web-based intervention manual from the original Dutch Version, the adaptation and implementation of all necessary technical and research-administrative requirements to successfully conduct the web-based randomized controlled trial and the evidence-based training of all study therapists including the implementation of therapists supervision. The investigators further assess adherence of the patients and therapists, the response rate and the patient satisfaction. Furthermore, preliminary efficacy of the intervention will be tested assessing levels of fatigue and quality of life at each measurement point.

Study Design: The design of this pilot web-based intervention on treating fatigue will be a non-randomised prospective non-controlled before-and-after study, in which observations will be made only in a patient group that receives the intervention. No control group will be recruited. Assessments will be conducted on the three measurement points: before the therapy (T0), after the intervention (T1) and 3 months after the intervention (T2).

Intervention: The internet-based cognitive behavioral therapy on postcancer fatigue includes two face-to-face sessions with their therapist and eight web-based treatment modules, each approximately 45 minutes in length, delivered over 6 months. The intervention will be specifically tailored to the individual needs of each patient: The therapy model of cancer-related fatigue distinguishes six perpetuating factors: 1) insufficient processing of being diagnosed with Hodgkin lymphoma and being treated for it; 2) excessive fear of disease recurrence; 3) inactivity or a dysregulated (physical) activity pattern; 4) dysfunctional fatigue-related beliefs; 5) dysregulated sleep-wake pattern and 6) lack of social support. For each of these six cognitive-behavioural factors that can perpetuate fatigue a treatment module has been developed. The intervention will consist of a maximum of eight treatment modules: aside from the six modules addressing the fatigue maintaining factor there is a module on goal formulation and realization of goals.

Recruitment: the recruitment will be realized on the basis of two ongoing trials of the German Hodgkin study group (HD 16- HD18) where fatigue of the patients is measured continuously.

Duration: The duration for patients will be 9 months (6 months intervention, 3 month-follow-up assessment). The duration of the whole study will be 18 months.

ELIGIBILITY:
Inclusion Criteria:

* fluency in German language
* able to access the internet and use and follow a web-based Cognitive Behavioral intervention
* in complete remission after treatment for newly diagnosed HL without signs of relapse (no previous relapse)
* clinically relevant fatigue symptoms enduring at least 12 months after end of treatment (QLQ-C30 FA-12 ≥ 30 over at least two time points within the previous assessments in the course of the GHSG-trials)
* fatigue being related to HL and its treatment and interferes with usual functioning, i.e. fulfills the definition of CRF [1, 16].

Exclusion Criteria:

* Major communication difficulties
* severe cognitive impairment that would interfere with a patient's ability to give informed consent for research (indicated by the medical care team)
* Karnofsky Performance Status scale score < 70 predicting an expected survival of less than 6 months
* somatic co-morbidities that could explain the presence of severe fatigue (e.g. Chronic Obstructive Pulmonary Disease or heart failure) according to the hemato-oncologists examining the potential participant before inclusion for the study
* history of relapsed or refractory HL
* clinical symptoms which may indicate a relapse of HL
* current depressive disorder and related psychotropic or psychological treatment
* Currently receiving medical and/or psychological treatment for a psychiatric disorder, other than the use of an anti-depressant
* current treatment aimed at fatigue
* previous attempt to treat fatigue with behavioral psychological therapy
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Response rate | The assessment period for this outcome will be from the start of recruitment until the inclusion of the last patient, which will be about 1 year.
  The investigators will assess the amount of eligible patients which are willing to participate in the study relative to the amount of patients who were invited to participate.
Patient adherence | During the intervention phase for each patient, which will be about sixth months.
  Patient adherence will be assessed via documentation of patient drop-outs. In detail, we will document whether patients leave the study during the treatment (and if yes, at what stage).
Patient satisfaction | Assessed only once for each patient, immediately after the patient has completed the intervention.
  Assessed by a questionnaire (Working Alliance Inventory - short form revised). The total sum score across the 12 items, rated on a five-point Likert scale, will be presented (ranging from 12 to 60). Higher values present higher satisfaction.
Therapist adherence | Assessed during the intervention phase for each patient, i.e., within about 6 six months.
  Using information of the therapy protocols of each participant, it will be assessed if the treatment sessions were done according to the treatment protocol.

SECONDARY OUTCOMES:
Levels of fatigue 1 | Assessed at three time points: before the intervention, immediately after the intervention and 3 months after the intervention
  Assessed by a questionnaire, the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Module Measuring Cancer-Related Fatigue (EORTC QLQ-FA12). The questionnaire assesses the level of cancer-related fatigue. The sum score across all 12 items, rated on a 4-point Likert scale, will be reported (total range: 12-48). Higher values indicate higher levels of fatigue (i.e., higher values indicate a worse outcome).
Levels of fatigue 2 | Assessed at three time points: before the intervention, immediately after the intervention and 3 months after the intervention
  Levels of fatigue will additionally assessed by a second questionnaire, the Checklist Individual Strength - Subscale Fatigue Severity. The scale assesses the level of cancer-related fatigue. The sum score across all 8 items, rated on a 7-point Likert scale, will be presented (total range: 8 - 56). Higher values indicate higher levels of fatigue (i.e., higher values indicate a worse outcome).
Global quality of life | Assessed at three time points: before the intervention, immediately after the intervention and 3 months after the intervention
  Global quality of Life will be assessed by the European Organisation for Research and Treatment of Cancer (EORTC), Quality of Life-questionnaire (EORTC QLQ-C30). Global quality of life is assessed in a 2-item subscale of the questionnaire, each rated on a 7-point-Likert scale (total range: 2-14). According to the questionnaire manual, however, the sum score of the two items will be linear-transformed to a 0-100 scale, with higher values indicating higher levels of quality of life (i.e., higher values indicate a better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mehnert, Prof. Dr., Principal Investigator — University of Leipzig; Peter Borchmann, Prof. Dr., Principal Investigator — University of Cologne
Locations (2):
- Germany (2):
  - University Medical Center Leipzig, Leipzig, Saxony
  - University Medical Center Cologne, Cologne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esser P, Muller H, Borchmann P, Kreissl S, Knoop H, Platzbecker U, Vucinic V, Mehnert-Theuerkauf A. Web-Based Cognitive-Behavioral Therapy to Reduce Severe Cancer-Related Fatigue Among Survivors of Hodgkin Lymphoma: A Feasibility Study. J Clin Psychol Med Settings. 2023 Dec;30(4):856-865. doi: 10.1007/s10880-023-09944-6. Epub 2023 Feb 20. PMID 36808045